CLINICAL TRIAL: NCT00617409
Title: A Randomized Phase II Trial Using Dendritic Cells Transduced With an Adenoviral Vector Containing the p53 Gene to Immunize Patients With Extensive Stage Small Cell Lung Cancer in Combination With Chemotherapy With or Without All Trans Retinoic Acid
Brief Title: To Immunize Patients With Extensive Stage SCLC Combined With Chemo With or Without All Trans Retinoic Acid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15206; 105790 (Other: USF IRB); 0147NE (Other: IBC); 0705-857 (Other: OBA); NCT00618891 (obsolete NCT alias)
Record Dates: First submitted 2008-02-05; First posted 2008-02-18 (Estimated); Results first posted 2016-11-01 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Small Cell Lung Cancer
Keywords: SCLC; vaccine; immunize
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Paclitaxel; Antineoplastic Agents; Drug Therapy; INGN 225; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard of Care (Active Comparator): Arm A - Active Comparator: Observation (Standard of Care) + Second Line Chemotherapy
  Interventions: Drug: Paclitaxel
- Ad.p53-DC Vaccines (Experimental): Arm B - Experimental: Ad.p53-DC vaccines + Second Line Chemotherapy
  Interventions: Drug: Paclitaxel; Biological: Drug: Ad.p53-DC vaccines
- Ad.p53-DC Vaccines + ATRA (Experimental): Arm C - Experimental: Ad.p53-DC vaccines + All -trans Retinoic Acid (ATRA) + Second Line Chemotherapy
  Interventions: Drug: Paclitaxel; Biological: Drug: Ad.p53-DC vaccines; Drug: All -trans Retinoic Acid (ATRA)

INTERVENTIONS:
Drug: Paclitaxel — All groups wil receive paclitaxel as second line chemotherapy if their cancer spreads. At any point when a patient develops evidence of progressive disease, the patient will be treated with second-line chemotherapy. Paclitaxel will be given at a dose of 200 mg/m² on day 1 of 21 day cycles.
  Other Names: Antitumor agent; Chemotherapy
Biological: Drug: Ad.p53-DC vaccines — Patients randomized to Arm B will receive vaccinations on 3 occasions, at 2 week intervals. 1-5x106 p53 positive DCs in 1 ml will be injected intradermally into 4 separate sites (0.25 ml injected at each site), in bilateral proximal upper and lower extremities (in the regions of the axillary and inguinal nodal basins). Patients will be restaged approximately 2-3 weeks after vaccine # 3 (first vaccine course). If patients show no sign of disease progression at restaging, then a second leukopheresis will be performed. Patients will then be vaccinated 3 more times (second vaccine course) at 4-week intervals, for a total of 6 possible vaccines. Restaging will occur 2-4 weeks after completing the second vaccine course. Patients in Arm C will receive vaccines at the same dose and schedule as described for patients in Arm B. In addition, they will receive 150 mg/m² of ATRA for 3 days prior to each vaccine administration (followed by vaccine administration on the fourth day).
  Other Names: INGN 225
  Arms: Ad.p53-DC Vaccines; Ad.p53-DC Vaccines + ATRA
Drug: All -trans Retinoic Acid (ATRA) — The patients in Arm C will receive vaccines at the same dose and schedule as described for patients in Arm B. In addition, they will receive 150 mg/m² of ATRA for 3 days prior to each vaccine administration (followed by vaccine administration on the fourth day).
  Other Names: tretinoin; Vesanoid; INGN 225
  Arms: Ad.p53-DC Vaccines + ATRA

SUMMARY:
The purpose of this research study is to test a tumor (cancer) vaccine given along with chemotherapy to determine if this vaccine will increase the chances of the tumor shrinking and/or the amount of time that people who have this disease will live.

DETAILED DESCRIPTION:
After initial diagnosis patients will be treated with a standard platinum/etoposide regimen. This standard first-line chemotherapy may/will be administered to patients under the direction of their primary medical oncologist inside or outside of the Moffitt Cancer Center. Patients will receive the platinum drug on day 1 and etoposide on days 1-3 of each 21-day cycle for 4-6 cycles. Patients who have progressive disease (PD) at this point are changed to second line chemotherapy, and will not be eligible to participate in this clinical trial. Patients who achieve a complete response (CR), partial response (PR), or stable disease (SD) after standard first-line chemotherapy will be enrolled. Radiographic studies and tumor measurements are repeated 3-6 weeks after the last dose of chemotherapy (+/- PCI) and may be repeated after prophylactic cranial irradiation (PCI) at the discretion of the principal investigator (PI) and treating physician.

PCI will be permitted at the discretion of the treating oncologist(s). The initial radiation consultation and simulation should occur as soon as the final staging has occurred. Ideally, treatment should commence 1-2 weeks after final staging has been confirmed and will be administered in 10-15 fractions over a 2-3 week period, as recommended by the treating radiation oncologist. Although steroid use is not prohibited, it is recommended and preferred that they not be used during PCI (steroids will have to be discontinued ≥ 2 weeks before first vaccination). PCI can also be considered between vaccines #4 and #5 or vaccine #5 and #6 in those patients eligible for the second course of vaccinations. Systemic dose of steroids will NOT be allowed in these cases unless strictly necessary and after discussion with the PI.

Patients who achieve CR, PR or SD after the completion of first line chemotherapy +/- PCI will be screened for initial registration. Screening tests and procedures will be performed approximately 4-6 weeks after the completion of first line chemotherapy or 6-9 weeks after completion of PCI. Ideally, screening should be completed 1-2 weeks prior to leukopheresis.

Patients who successfully complete the screening exams for initial registration will be randomized into one of three study arms.

ELIGIBILITY:
Inclusion Criteria at the time of initial registration:

* Patients must have a histological confirmed diagnosis of Small Cell Lung Cancer (SCLC)
* Must have extensive stage SCLC
* Must have completed first line chemotherapy: 4-6 cycles of a standard platinum/etoposide regimen and PCI if chosen at the discretion of the treating Oncologist
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Acceptable (adequate) organ function including:

  * White blood count (WBC) >2,500/mm³ and Absolute neutrophil count (ANC) >1,200/mm³
  * Platelets > 75,000/mm³
  * Hematocrit > 24% OR Hemoglobin ≥8.5g/dl
  * Bilirubin < 2.0 mg/dl
  * Creatinine < 2.0 mg/dl
  * Aspartic transaminase (AST/SGOT) ≤2 x upper limit of normal (ULN)
  * Alkaline phosphatase ≤3 x ULN
* Patients must have achieved responsive or non-progressive disease status (stable disease [SD], partial response [PR], or complete response [CR]) assessed 4-6 weeks after the last cycle of first line chemotherapy. SD, PR or CR may be confirmed after completion of prophylactic cranial irradiation (PCI) at the discretion of the principal investigator (PI) after discussion with the treating oncologist.
* Males and Females of reproductive potential must agree to use effective contraception during the study and for at least 4 weeks after the last dose of ATRA. Patients are instructed and agree to notify the principal investigator should a pregnancy occur for themselves or their partner.
* Willing and able to sign written informed consent and be able to comply with the study protocol for the duration of the study

Exclusion Criteria at the time of initial registration:

* Patients with severe, uncontrolled intercurrent illness or infection
* Anticipated requirement for systemic chronic steroid use at the time of vaccination, unless specifically indicated for dose supplementation or replacement of established corticosteroid insufficiency
* Receiving systemic doses of corticosteroids should have them discontinued ≥ 2 weeks prior to starting vaccination (this include patients receiving steroids with PCI). Inhaled steroids should also be discontinued if at all possible. Chronic, stable doses of inhaled steroids for the treatment of chronic obstructive pulmonary disease (COPD), etc. are allowed if in the opinion of the treating physician(s) they cannot be stopped.
* Any pre-existing immunodeficiency condition, or a known history of human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C
* Uncontrolled and/or symptomatic central nervous system (CNS) metastasis
* Pregnant or lactating women. A pregnancy test-serum Beta human chorionic gonadotropin (bHCG) will be obtained during the screening process.
* Have received any chemotherapy other than the first line chemotherapy specified in the study protocol: standard platinum/etoposide regimen
* Have received any prior investigational drugs including immunotherapy, gene therapy, hormone therapy, biologic therapy for treatment of SCLC
* Any known pre-existing autoimmune disorder
* History of a second malignancy within the previous 3 years. Exceptions include: non-melanoma skin cancers, any in-situ carcinomas and successfully treated early stage malignancies without evidence of recurrence for > 18 months.
* Have not recovered from any chemotherapy-related or other therapy-related toxicity at study entry
* Have had major surgery without full recovery or major surgery within 3 weeks of the start of vaccine treatment
* Patients with other significant diseases or disorders that, in the Investigator's opinion, would exclude them from the study

Pre-Pheresis Criteria:

* Patients must have had a successful harvest of peripheral blood mononuclear cell (PBMC) with leukopheresis at least 6-10 weeks after chemotherapy.
* ECOG performance status of 0-2
* The last dose of first line chemotherapy must have been administered at least 4 weeks prior to the first vaccine administration.
* Patients who received radiation therapy: last dose of radiation must have been completed at least 2 weeks prior to the first vaccine administration and the patient must have recovered from the toxic effects of the treatment prior to study enrollment (except for alopecia)
* Patients who received steroid therapy: last steroid dose must have been given at least 2 weeks prior to the first vaccine administration
* Adequate organ function:

  * WBC > 2,500/mm³ and ANC >1,200/mm³
  * Platelets > 75,000/mm³
  * Hematocrit > 25%
  * Hemoglobin ≥9g/dl
  * Bilirubin < 2.0 mg/dl
  * Creatinine < 2.0 mg/dL
  * AST/SGOT ≤ 2 x ULN
  * Alkaline phosphatase < 3 x ULN
* Patients must have signed informed consent at initial registration.
* HLA-A*0201 Testing as determined by flow cytometry followed by molecular analysis of a peripheral blood specimen, however this result will not be an inclusion criterion

Pre-Paclitaxel Eligibility:

* Progressive disease after observation (Arm A) or vaccinations (Arms B and C)
* ECOG performance status of 0-2
* Adequate organ function:

  * WBC > 2,500/mm³ and ANC >1,200/mm³
  * Platelets > 75,000/mm³
  * Hematocrit > 25%
  * Hemoglobin ≥9g/dl
  * Bilirubin < 2.0 mg/dl
  * Creatinine < 2.0 mg/dL
  * AST/SGOT ≤ 2 x ULN
  * Alkaline phosphatase < 3 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2007-10-02 (Actual); Primary Completion 2015-09-21 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Antonia, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ad.p53-DC Vaccines + ATRA: Arm C - Experimental: Ad.p53-DC vaccines + All -trans Retinoic Acid (ATRA) + Second Line Chemo
Period: Overall Study
Arm/Group | Standard of Care | Ad.p53-DC Vaccines | Ad.p53-DC Vaccines + ATRA
Started | 18 | 20 | 31
Completed | 2 | 2 | 4
Not Completed | 16 | 18 | 27
Not completed — Withdrawal by Subject | 4 | 1 | 2
Not completed — Adverse Event | 0 | 2 | 3
Not completed — Disease Progression | 8 | 8 | 18
Not completed — Death | 3 | 5 | 4
Not completed — Alternative Therapy | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All participants.
Groups:
- Arm A - Active Comparator: Active Comparator: Observation (Standard of Care) + Second Line Chemotherapy
- Arm B - Experimental: Experimental: Ad.p53-DC vaccines + Second Line Chemotherapy
- Arm C - Experimental: Experimental: Ad.p53-DC vaccines + ATRA + Second Line Chemo
- Total: Total of all reporting groups
Arm/Group | Arm A - Active Comparator | Arm B - Experimental | Arm C - Experimental | Total
Number analyzed (Participants) | 18 | 20 | 31 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 19 | 41
  >=65 years | 8 | 8 | 12 | 28
Age, Continuous [Mean (Full Range); unit: years] | 63 [44 to 74] | 63 [52 to 75] | 62.45 [49 to 78] | 62.75 [44 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 16 | 36
  Male | 11 | 7 | 15 | 33
Region of Enrollment [Number; unit: participants]
  United States | 18 | 20 | 31 | 69

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate (RR)
Description: Overall Response: Complete Response (CR) + Partial Response (PR) + Stable Disease (SD). Efficacy of second line chemotherapy (single agent paclitaxel) after progression following the dendritic cell(DC)-based p53 vaccine (Ad.p53-DC vaccine), with (Arm C). To estimate the objective tumor response rate for each treatment group. Tumor response to be assessed via radiographic imaging after every 2 cycles of chemotherapy (paclitaxel). CR: Disappearance of all target lesions. PR: At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease (PD), taking as reference the smallest sum LD since the treatment started. PD: At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 12 months
Population: All participants.
Measure: Number; unit: participants
Arm/Group | Standard of Care | Ad.p53-DC Vaccines | Ad.p53-DC Vaccines + ATRA
Number analyzed (Participants) | 18 | 20 | 31
participants
  Overall Response | 8 | 6 | 12
  Progressive Disease | 1 | 5 | 6

2. Secondary Outcome: Overall Survival (OS)
Description: To evaluate the survival of all patients enrolled on an intent-to-treat basis. Overall survival per treatment arm.
Time Frame: Up to 24 months
Population: All participants.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Ad.p53-DC Vaccines + ATRA: Arm C - Experimental: Ad.p53-DC vaccines + ATRA + Second Line Chemo
Arm/Group | Standard of Care | Ad.p53-DC Vaccines | Ad.p53-DC Vaccines + ATRA
Number analyzed (Participants) | 18 | 20 | 31
months | 12.17 [9.27 to 18.83] | 6.32 [5.13 to 13.93] | 6.20 [4.17 to 11.57]

ADVERSE EVENTS:
Time Frame: 6 years, 6 months
Arm/Group | Arm A - Active Comparator | Arm B - Experimental | Arm C - Experimental
Serious Adverse Events (participants affected / at risk) | 7/18 | 9/20 | 12/31
Other Adverse Events (participants affected / at risk) | 16/18 | 17/20 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Active Comparator (N=18) | Arm B - Experimental (N=20) | Arm C - Experimental (N=31)
Blood and lymphatic system disorders - Other, Leukopenia/Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac ischemia/infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Death NOS (General disorders) | 0 (0) | 3 (3) | 5 (5)
Fever (in the absence of neutropenia) (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain - Chest wall (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain - Chest/thorax NOS (General disorders) | 0 (0) | 1 (1) | 0 (0)
Rigors/chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutopenia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Infection with Grade 3 or 4 neutrophils - Mucosa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Leukocytes (total WBC) - low (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelets - low (Investigations) | 0 (0) | 0 (0) | 1 (1)
Pain - Bone (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pain - Head/headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (7) | 3 (3)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary/Upper Respiratory - Other, COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0)
Pulmonary/Upper Respiratory - Other, Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vessel injury-artery - Other NOS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Active Comparator (N=18) | Arm B - Experimental (N=20) | Arm C - Experimental (N=31)
Edema: limb (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Hemolysis (e.g., immune hemolytic anemia, drugrelated hemolysis) (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
Leukocytes (total WBC) - Low (Blood and lymphatic system disorders) | 1 (1) | 2 (6) | 5 (11)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (9)
Neutrophils/granulocytes (ANC/AGC) - Low (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Auditory/Ear - Other, Hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular/Visual - Other, Keratotic lesion-left side (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular/Visual - Other, Right sided ptosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision-blurred vision (Eye disorders) | 1 (1) | 2 (2) | 2 (2)
Anorexia (Gastrointestinal disorders) | 7 (11) | 5 (6) | 12 (15)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4) | 5 (6)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (3) | 2 (2) | 9 (10)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (3) | 0 (0) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Flatulance (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal - Other, Decrease color in stools (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal - Other, GI virus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal - Other, Increased burping (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 2 (2)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 3 (3) | 14 (22)
Pain - Absomen NOS (Gastrointestinal disorders) | 1 (1) | 2 (3) | 4 (5)
Pain - Esophagus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pain - Other, Pain at distal margins (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain - Stomach (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (3) | 1 (1) | 9 (13)
Fatigue (General disorders) | 8 (12) | 13 (19) | 22 (29)
Fever (in the absence of neutropenia) (General disorders) | 2 (2) | 1 (1) | 1 (1)
Flu-like syndrome (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pain - Chest/thorax NOS (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pain - Face (General disorders) | 0 (0) | 0 (0) | 2 (4)
Pain - Other, Upper quadrant (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain - Pain NOS (General disorders) | 0 (0) | 1 (1) | 0 (0)
Rigors/chills (General disorders) | 1 (1) | 1 (1) | 0 (0)
Sweating (diaphoresis) (General disorders) | 1 (1) | 2 (2) | 2 (3)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 1 (1) | 0 (0) | 3 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Bilirubin (hyperbilirubinemia) (Investigations) | 0 (0) | 0 (0) | 2 (2)
Creatinine - High (Investigations) | 0 (0) | 1 (1) | 2 (2)
Hemoglobin - Low (Investigations) | 3 (3) | 4 (5) | 6 (15)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Metabolic/Laboratory - Other, Elevated AST (Investigations) | 2 (2) | 0 (0) | 3 (3)
Platelets - Low (Investigations) | 1 (1) | 3 (3) | 6 (14)
Weight loss (Investigations) | 4 (4) | 1 (1) | 3 (3)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 4 (7)
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) - High (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (5)
Amylase (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 8 (18)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 5 (8)
Metabolic/Laboratory - Other, Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic/Laboratory - Other, Decreased HDL (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic/Laboratory - Other, Decreased protein (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic/Laboratory - Other, High total protein (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic/Laboratory - Other, Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolic/Laboratory - Other, Increased ALT (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (2)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (3)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 6 (9)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extraocular (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremitylower (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Pain - Back (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (7) | 5 (5)
Pain - Bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 7 (10)
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 2 (2)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (3) | 5 (8)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 4 (4)
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 6 (6)
Pain - Other, Flank (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain - Other, Hip (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain - Other, Rib/Rib cage (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Pain - Other, Shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3)
Ataxia (incoordination) (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1) | 3 (3)
Memory Impairment (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Neurology - Other, Numbness in lower legs and feet (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Neuropathy: cranial - CN IX Motor-pharynx; Sensory-ear, pharynx, tongue (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Neuropathy: cranial - CN VIII Hearing and balance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 3 (4) | 3 (4) | 9 (14)
Pain - Head/headache (Nervous system disorders) | 3 (4) | 4 (4) | 22 (65)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 2 (2) | 4 (5)
Mental status (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mood alteration - Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1)
Mood alteration - Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Incontinence, urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Obstruction, GU - Ureter (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urine color change (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pain - Breast (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pain - Pelvis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 9 (10) | 11 (16)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 11 (17) | 14 (20)
Hemorrhage/Bleeding - Other, Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pain - Pleura (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary/Upper Respiratory - Other, Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary/Upper Respiratory - Other, Absent breath sounds-right base (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary/Upper Respiratory - Other, Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatology/Skin - Other, erythema- chest wall and scalp (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatology/Skin - Other, Tightness of skin on hands (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 6 (11)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 3 (5) | 3 (4) | 7 (11)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 4 (4)
Pain - Scalp (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 5 (6)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (4)
Rash: dermatitis associated with radiation - Chemoradiation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash: dermatitis associated with radiation - Radiation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vascular - Other, Chronic venous stasis in legs (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Protocol V.10.1, 04/11/2012: Arm A was closed due to lack of feasibility; Arm B was closed at the end of the first stage due to lack of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes